CLINICAL TRIAL: NCT02723838
Title: A Phase 1b Study of Intratumoral REOLYSIN® in Combination With Gemcitabine and Cisplatin as Neoadjuvant Therapy in Muscle-invasive Transitional Cell Carcinoma of the Bladder
Brief Title: Study of Intratumoral REOLYSIN® in Combination With Gemcitabine and Cisplatin as Neoadjuvant Therapy in Muscle-invasive Transitional Cell Carcinoma of the Bladder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company has reprioritized clinical plans to focus on later-stage studies.
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 023
Record Dates: First submitted 2016-03-24; First posted 2016-03-31 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Muscle-invasive Transitional Cell Carcinoma of the Bladder
Keywords: Bladder; Cancer; REOLYSIN®; Gemcitabine; Cisplatin; Reovirus; Oncolytic virus
MeSH Terms: conditions — Neoplasms | interventions — reolysin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: REOLYSIN® — 3 cycles (each cycle = 21 days). Cohort 1: 3x10E10 TCID50 intratumoral via cystoscopy on Day 1 of each cycle. Cohort 2: 3x10E10 TCID50 intratumoral via cystoscopy on Day 2 of each cycle.
Drug: Gemcitabine — 3 cycles (each cycle = 21 days). Cohort 1: 1000mg/m2 intravenously on Day 2 and Day 9 of Cycle 2 and Cycle 3. Cohort 2: 1000mg/m2 intravenously on Day 1 and Day 8 of each cycle.
Drug: Cisplatin — 3 cycles (each cycle = 21 days). Cohort 1: 70 mg/m2 intravenously on Day 2 of Cycle 2 and Cycle 3. Cohort 2: 70 mg/m2 intravenously on Day 1 of each cycle.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of intratumoral REOLYSIN® therapy alone and in combination with standard neoadjuvant gemcitabine and cisplatin in muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
Reovirus Serotype 3 - Dearing Strain (REOLYSIN®) is a naturally occurring, ubiquitous, non-enveloped human reovirus. Reovirus has been shown to replicate selectively in Ras-transformed cells causing cell lysis. Activating mutations in Ras or mutations in oncogenes signaling through the Ras pathway may occur in as many as 80% of human tumors. The specificity of the reovirus for Ras-transformed cells, coupled with its relatively nonpathogenic nature in humans, makes it an attractive anti-cancer therapy candidate.

This is an open-label study of intratumoral REOLYSIN® in combination with standard of care neoadjuvant cisplatin/gemcitabine in patients with histologically and clinically confirmed muscle-invasive bladder cancer (T2-4) with or without pelvic lymph node involvement (N1-2) in Stage III and IV with no distant metastases (M0) and no prior systemic therapy for bladder cancer.

Treatment with intratumoral REOLYSIN® and chemotherapy is planned for 3 cycles followed by radical cystectomy or until unacceptable toxicity or another discontinuation criterion is met.

Two sequential treatment cohorts will be enrolled.

Patients in Cohort 1 will receive intratumoral REOLYSIN® on Cycle 1 Day 1, then 7-14 days later patients will receive intratumoral REOLYSIN® on Cycle 2 Day 1 plus intravenous neoadjuvant chemotherapy for 2 cycles (every 3 weeks) starting from Cycle 2 Day 2 followed by radical cystectomy. Three patients will be enrolled in this cohort. If there is a Dose Limiting Toxicity the cohort will be expanded to an additional 3 patients.

Upon completion of Cohort 1, Cohort 2 will be open to enrollment of 3 patients to receive 3 cycles of standard neoadjuvant chemotherapy on Day 1 and Day 8 of each cycle and intratumoral REOLYSIN® on Day 2 of each cycle (every 3 weeks). If there is a Dose Limiting Toxicity the cohort will be expanded to an additional 3 patients.

An Expansion Cohort will follow with up to 12 patients to be enrolled following either Cohort 1 or Cohort 2 treatment regimen based on the results of Cohort 1 and Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and clinically confirmed muscle-invasive bladder cancer (T2-4) with or without pelvic lymph nodes involvement (N1-2) in Stage III and IV (M0).
* ECOG performance status ≤2.
* Adequate liver function with a bilirubin within normal limits. Transaminases up to 3 x ULN (Grade 1) and alkaline phosphatase may be up to 2.5 x ULN (Grade 1).
* Adequate bone marrow function, as defined by neutrophils count of ≥1,500/mm3, and platelet count ≥100,000/ mm3.
* Adequate renal function (serum creatinine ≤1.5 times the ULN).
* Negative pregnancy test and reliable and appropriate contraceptive method during the study for a woman of childbearing potential. All female patients of childbearing age and all male patients with partners of childbearing age should use a reliable method of contraception, such as the barrier method, throughout the study and for 60 days after last treatment.
* Informed of the investigational nature of this study and must sign a written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Received any prior therapy for invasive bladder cancer including surgery, radiation therapy, chemotherapy or any other systemic anti-cancer therapy (prior intravesical therapy for non-invasive bladder cancer is acceptable including intravesical BCG and/or mitomycin and interferon).
* Evidence of lymph nodes or other metastatic disease beyond the pelvis (N3 and/or M1).
* Pre-existing immunosuppressive or connective tissue disorders that require immune suppressive drugs.
* History of HIV or active hepatitis.
* Any serious concurrent illness including; but not limited to, unstable angina pectoris, uncompensated congestive cardiac failure; myocardial infarct in the previous 6 months; cardiac arrhythmias or psychiatric illness that would limit compliance with study requirements.
* Pregnant or lactating.
* A history of hypersensitivity to gemcitabine and cisplatin or any component of the formulation.
* A prior malignancy, other than non-melanoma skin cancer, unless they have completed therapy at least 5 years prior to start of study and have no evidence of recurrent or residual disease.
* Unwilling or unable to sign informed consent document.
* In social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-28 (Estimated); Primary Completion 2017-09-30 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | During treatment and up to 28 days after treatment
  Nature, frequency, severity and timing of Adverse Events.
Pre- and post-treatment biopsies will be evaluated for tumor viability, percentage of necrosis, reovirus replication and tumor infiltration of immune cells and expression of PD-1 and PD-L1 | Assessed at surgery conducted following 3 3-week study treatment cycles

SECONDARY OUTCOMES:
Time to Treatment Failure (TTF) | By medical chart review until disease reoccurrence or 2 years from surgery, whichever occurs first first.
Disease Free Survival (DFS) | By medical chart review until disease reoccurrence or death or 2 years from surgery, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No